CLINICAL TRIAL: NCT06076733
Title: To Explore the Intervention Effect of High Definition-transcranial Alternating Current Stimulation (HD-tACS) on Consciousness Promotion in Patients With Chronic Consciousness Disorders and the Potential Neural Mechanism
Brief Title: Intervention Effect of Transcranial Alternating Current Stimulation (tACS) on Disorder of Consciousness (DOC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tACS-DOC
Record Dates: First submitted 2023-10-02; First posted 2023-10-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Disorders of Consciousness
Keywords: DOC tACS
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active group (Experimental): Twenty 2-mA sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes per session, twice daily over 10 consecutive days, and the stimulus frequency was set as 6Hz.
  Interventions: Device: high definition-transcranial alternating current stimulation
- sham group (Sham Comparator): Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Interventions: Device: sham transcranial alternating current stimulation

INTERVENTIONS:
Device: high definition-transcranial alternating current stimulation — tACS is described as a non-invasive form of brain stimulation that uses a low-intensity, alternating current applied directly to the head through scalp electrodes.
  Arms: active group
Device: sham transcranial alternating current stimulation — Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham group

SUMMARY:
To investigate the effect of high definition-transcranial alternating current stimulation(HD-tACS) on consciousness promotion in patients with chronic consciousness disorders and the underlying neural mechanism by EEG.

DETAILED DESCRIPTION:
Forty patients with chronic consciousness disorder who met the inclusion criteria were recruited with the informed consent of the family. All the participants were randomized to receive "active" or "sham" treatment protocol. Stimulation was performed using a alternating stimulator linked to one anodal electrode and four cathodal electrodes. The anodal electrode was placed over the left dorsolateral prefrontal cortex (DLPFC; F3 in the 10-20 international system of EEG placement), and the four cathodal electrodes (AFz, FCz, F7, and C5 in the 10-20 international system EEG placement) were placed around the anodal electrode to form a current loop. Twenty 2 milliampere (mA) sessions (ramp-up and ramp-down periods of 30 and 30 seconds, respectively) were applied for 20 minutes per session, twice daily over 10 consecutive days, and the stimulus frequency was set as 6 Hertz (Hz). Sham tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds. Before and after the tACS treatment, the state of consciousness was assessed according to coma recovery scale-revised(CRS-R), and19-channel EEG data were collected.

ELIGIBILITY:
Inclusion Criteria:

1. patients diagnosed as chronic disorders of consciousness based on CRS-R assessment by at least two professional neurologists;
2. the age requirement is between 18 and 75;
3. vital signs need to be stable;
4. no neuromuscular blockers and sedatives have been used within 24 hours before the study and the entire protocol;
5. no improvement in the state of consciousness was observed within one week before the start of the study.

Exclusion Criteria:

1. previous or current diagnosis of severe neurocognitive degenerative diseases;
2. metal implantation in the head;
3. previous surgical procedures resulted in skull defect;
4. previous history of epilepsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Coma Recovery Scale | Before intervention and one day after all intervention
  State of consciousness was assessed by two trained physicians in three different time periods using the Coma Recovery Scale-Revised (CRS-R), which has demonstrated good reliability and validity for the behavioral evaluation of disorder of consciousness (DOC) patients. Total score ranges from zero to twenty-three, with higher scores indicating better neurological function and prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Wang, PhD, Principal Investigator — Director of medical psychological department, Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China